CLINICAL TRIAL: NCT02322944
Title: China Patient-centered Evaluative Assessment of Cardiac Events II: Quality Improvement for Acute Myocardial Infarction
Brief Title: China PEACE II: Quality Improvement for Acute Myocardial Infarction
Acronym: PEACE-QI-AMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: MOST-2013BAI09B01
Record Dates: First submitted 2014-12-15; First posted 2014-12-23 (Estimated); Last update posted 2016-10-24 (Estimated); Status verified 2016-10

CONDITIONS: Acute Myocardial Infarction
Keywords: acute myocardial infarction; quality improvement; reperfusion therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Intervention group (Experimental): The intervention group will take the treatment quality improvement strategies and tools into implementation.
  Interventions: Behavioral: Quality improvement strategies and tools
- Control group (No Intervention): The control group will maintain the routine practice pattern.
- Process optimization group (Experimental): The process optimization group's clinical pathways and team building will be re-organized for the purpose of quality improvement, and develop individualized treatment strategies and process.
  Interventions: Behavioral: Quality improvement strategies and tools; Behavioral: Process optimization

INTERVENTIONS:
Behavioral: Quality improvement strategies and tools — Training in standardized treatment pattern; building quality management team and determining improvement goals; tools (a wristband in order to remind all medical staff involved in the treatment process; workflow posters and cards; a CRF including a flowchart to inform the management steps); periodical quality feedback report and regular quality meeting; study website serving as the communication platform.
  Arms: Intervention group; Process optimization group
Behavioral: Process optimization — Examining local hospitals' workflow to determine the key link affecting the rate of reperfusion therapy and its timeliness (such as thrombolytic drug preparation, cardiac catheterization laboratory preparation, transferring from the ER to the cath lab, interventional medical team gathering, etc.) and systems (such as pre-paid policy for thrombolysis or PPCI)
  Arms: Process optimization group

SUMMARY:
This study aims to develop quality improvement strategies and relevant tools focusing on reperfusion therapy in patients with STEMI, and to evaluate their effectiveness via a hospital-level cluster randomized clinical trial, based on the nationally representative collaborative network of over 100 hospitals established in China PEACE retrospective study. In a baseline survey period, through consecutively recruiting all eligible inpatients and collecting relevant medical information, the performance of all participating hospitals before the implementation of the intervention will be assessed. During the following intervention period, 6-10 hospitals that show the strong willingness and ability to collaborate will be selected as "process optimization group". Their clinical pathways and team building will be re-organized for the purpose of quality improvement, and develop individualized treatment strategies and process. Meanwhile, other participating hospitals will be divided into intervention and control groups in a 1:1 ratio, in which the intervention group will take the treatment improvement strategy into implementation, while the control group will maintain the routine practice pattern. All hospitals will consecutively recruit qualified patients in the same method adopted in baseline period. Then the reperfusion rates and other performance measures will be compared among different groups (process optimization, intervention and control).

DETAILED DESCRIPTION:
This study aims to develop quality improvement strategies and relevant tools focusing on reperfusion therapy in patients with STEMI, and to evaluate their effectiveness via a hospital-level cluster randomized clinical trial, based on the nationally representative collaborative network of over 100 hospitals established in China PEACE retrospective study. The primary outcome measure is reperfusion rate among eligible patients with STEMI, and secondary ones include timeliness of primary PCI (D2B) and fibrinolytic therapy (D2N). the assessment is based on consecutively recruiting all eligible inpatients, as well as collecting relevant medical information via a case report form finished by local doctors and central medical record abstraction.

During the first study period, the baseline performance of all 100 participating hospitals before the implementation of the intervention will be assessed.

During the following period, 3-5 PCI-capable and 3-5 non-PCI capable hospitals that show the strong willingness and ability to collaborate will be selected as "process optimization group". Their clinical pathways and team building will be re-organized for the purpose of quality improvement, and develop individualized treatment strategies and process, including examining local hospitals' workflow to determine the key link affecting the rate of reperfusion therapy and its timeliness (such as pre-paid policy for fibrinolytic or PPCI, thrombolytic drug preparation, cardiac catheterization laboratory preparation, transferring from the ER to the Cath lab, interventional medical team gathering, etc.). Also, QI strategies and tools developed in the current study will be provided to these hospital, including training in standardized treatment pattern; building quality management team and determining improvement goals; periodical quality feedback report and regular quality meeting; tools like a wristband in order to remind all medical staff involved in the treatment process, workflow posters and cards, a CRF including a flowchart to inform the management steps, study website serving as the communication platform.

Meanwhile, other participating hospitals will be divided into intervention and control groups in a 1:1 ratio using minimization allocation, in which the intervention group will take the QI strategies and tools developed in the current study as mentioned above, while the control group will maintain the routine practice pattern. Then the outcome measures and other performance indicators will be compared among different groups (process optimization, intervention and control).

ELIGIBILITY:
Inclusion Criteria:

* Patients with STEMI who arrive at the hospital within 12 hours from the symptoms onset.

Exclusion Criteria:

* Received reperfusionthrombolytic therapy before the index hospitalization;
* AMI occurring during hospitalization;
* Chest trauma resulting in secondary acute myocardial infarction.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8000 (Actual)
Dates: Start 2014-12; Primary Completion 2016-06 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Reperfusion therapy rate | 24 hours after admission
  Reperfusion therapy rate is defined as utilization rate of thrombolytic therapy or primary PCI treatment among patients indicated with the reperfusion therapy.

SECONDARY OUTCOMES:
Timeliness of primary PCI | 24 hours after admission
  The proportion of door to balloon (D2B) within 90 minutes among all patients receiving PPCI.
Timeliness of thrombolytic therapy | 24 hours after admission
  The proportion of door to needle time (D2N) within 30 minutes among all patients receiving fibrinolytic therapy.
Timeliness of primary PCI | 24 hours after admission
  Door to balloon (D2B) time
Timeliness of thrombolytic therapy | 24 hours after admission
  Door to needle (D2N) time

OTHER OUTCOMES:
In-hospital mortality | 10 days on average (during hospitalization)
  Proportion of in-hospital mortality or withdraw treatment due to a terminal status at discharge.
Aspirin use within 24 hours | 24 hours after admission
  Proportion of aspirin use within 24 hours of admission among eligible patients
Heparin use within 24 hours | 24 hours after admission
  Proportion of heparin use within 24 hours of admission among eligible patients
Evaluation of left ventricular function | 24 hours after admission
  Proportion of left ventricular function evaluation within 24 hours of admission among all patients.
β-blockers use during hospitalization | 10 days on average (during hospitalization)
  Proportion of β-blockers use during hospitalization among eligible patients.
Statins use during hospitalization | 10 days on average (during hospitalization)
  Proportion of statins use during hospitalization among eligible patients.
ACEI/ARB use during hospitalization | 10 days on average (during hospitalization)
  Proportion of ACEI/ARB use during hospitalization among eligible patients.
Aspirin use at discharge | 10 days on average (during hospitalization)
  Proportion of aspirin use at discharge among eligible patients.
Clopidogrel (or ticagrelor) use at discharge | 10 days on average (during hospitalization)
  Proportion of Clopidogrel (or ticagrelor) use at discharge among eligible patients.
β-blockers use at discharge | 10 days on average (during hospitalization)
  Proportion of β-blockers use at discharge among eligible patients.
ACEI/ARB use at discharge | 10 days on average (during hospitalization)
  Proportion of ACEI/ARB use at discharge among eligible patients.
Statins use at discharge | 10 days on average (during hospitalization)
  Proportion of statins use at discharge among eligible patients.

CONTACTS AND LOCATIONS:
Overall Officials: Lixin Jiang, MD, PhD, Principal Investigator — Fuwai Hospital, National Center for Cardiovascular Diseases
Locations (1):
- Qinyang People's Hospital, Jiaozuo, Henan, China